CLINICAL TRIAL: NCT06543654
Title: Evaluation of Template Assisted Monochromatic Structural Colored Versus Universal Multi-Shade Direct Composite Veneers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Abd El Ghany Mohammed, Assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Direct veneers
Record Dates: First submitted 2024-08-04; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Tooth Discoloration
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical study
Who Masked: Participant, Outcomes Assessor
Masking Description: This clinical trial was double-blind since the evaluators who were not included in the restorative procedures and the participants were blinded to tested groups, but the operator wasn't blinded to these groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omnichroma (Experimental): Monochromatic structural colored composite
  Interventions: Other: Omnichroma; Other: Ceram. X Spectra
- Ceram. X Spectra (Experimental): Universal multi shade composite
  Interventions: Other: Omnichroma; Other: Ceram. X Spectra

INTERVENTIONS:
Other: Omnichroma — Each participants had two kinds of veneers
Other: Ceram. X Spectra — Ceram. X Spectra

SUMMARY:
The aim of this study was to conduct a clinical trial utilizing a modified split-mouth, double-blinded, randomized strategy to clinically assess template assisted one shade structural colored versus universal multi-shade direct composite veneers

DETAILED DESCRIPTION:
The superior mechanical qualities, superb aesthetics, and versatility of resin-based composites (RBCs) make them popular choices for direct restorative applications. Compared to their predecessors, nanocomposites have shown superior qualities since nanotechnology was introduced in the production of dental RBCs.

A restoration's aesthetic integration is mostly the result of its chromatic characteristics. Pigments included in the composition of the restorative material typically control the selective reflection of wavelengths to emulate the natural tooth. In order to better reflect the broad color range that characterizes real dentition, RBCs have more recently employed the phenomena of "structural color" .

Thanks to the novel property of resins, color differences between the tooth and the restoration are eliminated or balanced out as perceived color of a region moves toward the color of the surrounding area . Additionally, as opposed to multi-shade RBCs, single-shade RBCs eliminate the need to select between various resin shades, streamlining the color choosing procedure and cutting down on time lost during the clinical resin selection process. The Vita Classic Shade Guide's shades can all be matched with these materials.

ELIGIBILITY:
Inclusion Criteria:

* better dental hygiene
* discolored vital anterior teeth

Exclusion Criteria:

* Para functional activities
* Non-vital teeth

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation was performed at baseline, six, nine, twelve, and eighteen months by two calibrated examiners using modified United States Public Health Service (USPHS) criteria | eighteen months
  The perfect clinical scenario was represented by a score of 0, clinically acceptable by a score of 1, dubious by a score of 2, and clinically unsatisfactory by a score of 3 and 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kobayashi S, Nakajima M, Furusawa K, Tichy A, Hosaka K, Tagami J. Color adjustment potential of single-shade resin composite to various-shade human teeth: Effect of structural color phenomenon. Dent Mater J. 2021 Jul 31;40(4):1033-1040. doi: 10.4012/dmj.2020-364. Epub 2021 Apr 20. PMID 33883353
- [Result] Arai Y, Kurokawa H, Takamizawa T, Tsujimoto A, Saegusa M, Yokoyama M, Miyazaki M. Evaluation of structural coloration of experimental flowable resin composites. J Esthet Restor Dent. 2021 Mar;33(2):284-293. doi: 10.1111/jerd.12674. Epub 2020 Oct 24. PMID 33098228
- [Result] Furusawa K, Kobayashi S, Yamashita A, Tichy A, Hosaka K, Shimada Y, Nakajima M. Effect of filler load on structural coloration and color adjustment potential of resin composites. Dent Mater J. 2023 May 30;42(3):343-350. doi: 10.4012/dmj.2022-199. Epub 2023 Jan 28. PMID 36709985
- [Result] Kam Hepdeniz O, Temel UB. Clinical survival of No-prep indirect composite laminate veneers: a 7-year prospective case series study. BMC Oral Health. 2023 May 3;23(1):257. doi: 10.1186/s12903-023-02949-5. PMID 37138297
- [Result] Castro FLA, Durand LB. Influence of cavity wall thickness on the color adjustment potential of single-shade resin composites. J Am Dent Assoc. 2024 Jul;155(7):605-613. doi: 10.1016/j.adaj.2024.03.006. Epub 2024 May 31. PMID 38819355
- [Result] Miranda AO, Favoreto MW, Matos TP, Castro AS, Kunz P, Souza JL, Carvalho P, Reis A, Loguercio AD. Color Match of a Universal-shade Composite Resin for Restoration of Non-carious Cervical Lesions: An Equivalence Randomized Clinical Trial. Oper Dent. 2024 Jan 1;49(1):20-33. doi: 10.2341/23-021-C. PMID 38057996